CLINICAL TRIAL: NCT01366547
Title: A Randomized, Open-Label, Single-Dose, 3-Period, Crossover Evaluation of the Relative Bioavailability of Two Experimental Fixed-Dose Combination Tablet Formulations of Dolutegravir 50 mg/Abacavir 600 mg/Lamivudine 300 mg Compared to Co-Administered Dolutegravir 50 mg and EPZICOM™ (Abacavir 600 mg/Lamivudine 300 mg) Tablets in Healthy Adult Subjects
Brief Title: Relative Bioavailability Study of Two New Dolutegravir/Abacavir/Lamivudine Fixed Dose Combination Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Cheri Hudson; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 114581
Record Dates: First submitted 2011-05-26; First posted 2011-06-06 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Healthy Subjects; Infection, Human Immunodeficiency Virus
Keywords: Bioavailability; Lamivudine; Dolutegravir; integrase; Abacavir
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; abacavir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Subjects will be randomized in a three-way crossover design to receive a single dose of each of two different tablet formulations of dolutegravir 50 mg/abacavir 600 mg/lamivudine 300 mg or dolutegravir 50 mg plus EPZICOM (abacavir 600mg/lamivudine 300 mg). There will be a screening visit within 30 days prior to first dose and a follow-up visit 7-14 days after the last dose.
  Interventions: Drug: Dolutegravir 50 mg/abacavir 600 mg/lamivudine 300 mg; Drug: Dolutegravir 50 mg; Drug: abacavir 600 mg/lamivudine 300 mg

INTERVENTIONS:
Drug: Dolutegravir 50 mg/abacavir 600 mg/lamivudine 300 mg — Dolutegravir 50 mg/abacavir 600 mg/lamivudine 300 mg is an experimental fixed dose combination tablet of an experimental integrase inhibitor (dolutegravir) and two FDA approved nucleoside reverse transcriptase inhibitors (abacavir and lamivudine)
Drug: Dolutegravir 50 mg — Dolutegravir is an experimental drug in the integrase inhibitor class that is being studied for the treatment of HIV infection.
Drug: abacavir 600 mg/lamivudine 300 mg — This is an FDA approved fixed dose combination tablet of two nucleoside reverse transcriptase inhibitors
  Other Names: KIVEXA. This is a trademark of ViiV Healthcare; EPZICOM. This is a trademark of ViiV Healthcare.

SUMMARY:
Dolutegravir (DTG, GSK1349572) is a next-generation integrase inhibitor (INI) currently in phase 3 clinical trials for human immunodeficiency virus (HIV). Fixed-dose combinations (FDCs) have greatly simplified the treatment of patients with HIV. While Atripla (an FDC of tenofovir (TDF), emtricitabine (FTC) and efavirenz (EFV)) has become the preferred first line regimen due in large part to its convenient presentation as a full treatment regimen in a single product, other options are needed. A fixed-dose combination of DTG/abacavir (ABC)/lamivudine (3TC) is one such opportunity.

This is a single-center, randomized, open-label, 3-period crossover study in healthy adult subjects to evaluate the single-dose relative bioavailability of two experimental oral DTG 50 mg/ABC 600 mg/3TC 300 mg FDC tablet formulations compared to co-administration of the separate tablet formulations (DTG 50 mg tablet and EPZICOM), with each dose administered in the fasted state. Approximately 18 subjects will be enrolled and randomized to one of 6 different treatment sequences. There will be a screening visit within 30 days prior to the first dose of study drug and a follow up visit within 7-14 days after the last dose. There will be a 7 day washout between doses in each treatment period.

The following PK parameters for DTG, ABC and 3TC will be measured: area under the concentration curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity)), Area under the concentration-time curve from time zero (pre-dose) to the time of the last quantifiable concentration (AUC (0-t)), maximum observed concentration (Cmax), lag time before observation of drug concentrations (tlag), time of occurrence of Cmax (tmax), terminal phase half-life (t½), apparent clearance following oral dosing (CL/F) and apparent terminal phase volume of distribution (Vz/F).

DETAILED DESCRIPTION:
Official Title - Randomized, Open-Label, Single Dose, 3 Period, Crossover Evaluation of the Relative Bioavailability of Two Experimental Fixed-Dose Combination Tablet Formulations of Dolutegravir 50 mg/Abacavir 600 mg/Lamivudine 300 mg Compared to Co administered Dolutegravir 50 mg and EPZICOM™ (Abacavir 600 mg/Lamivudine 300 mg) Tablets in Healthy Adult Subjects.

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential or child-bearing potential and agrees to use one of the contraception methods listed in the protocol until the follow-up visit.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol until 84 days after the last dose of study drug.
* Body weight greater than 50 kg for males and greater than 45 kg for females and BMI within the range 18.5- 31.0 kg/m2 (inclusive).
* ALT, alkaline phosphatase and bilirubin less than 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* A negative HLA-B*5701 allele screening assessment
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as:An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. 7. Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of Gilbert's disease.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening ECG outside of protocol limits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Plasma DTG AUC(0-infinity) | 48 hours post dose
Plasma ABC AUC(0-infinity) | 48 hours post dose
Plasma 3TC AUC(0-infinity) | 48 hours post dose
Plasma DTG AUC(0-t) | 48 hours post dose
Plasma ABC AUC(0-t) | 48 hours post dose
Plasma 3TC AUC(0-t) | 48 hours post dose
Plasma DTG Cmax | 48 hours post dose
Plasma ABC Cmax | 48 hours post dose
Plasma 3TC Cmax | 48 hours post dose

SECONDARY OUTCOMES:
Change from baseline in 12-lead ECG | 48 hours post dose
Plasma DTG tlag | 48 hours post dose
Number of subjects with adverse events | 48 hours post dose
Toxicity grading of clinical laboratory tests | 48 hours post dose
Change from baseline in vital signs (BP and HR) | 48 hours post dose
Plasma ABC tlag | 48 hours post dose
Plasma 3TC tlag | 48 hours post dose
Plasma DTG tmax | 48 hours post dose
Plasma ABC tmax | 48 hours post dose
Plasma 3TC tmax | 48 hours post dose
Plasma DTG t½ | 48 hours post dose
Plasma ABC t½ | 48 hours post dose
Plasma 3TC t½ | 48 hours post dose
Plasma DTG CL/F | 48 hours post dose
Plasma ABC CL/F | 48 hours post dose
Plasma 3TC CL/F | 48 hours post dose
Plasma DTG Vz/F | 48 hours post dose
Plasma ABC Vz/F | 48 hours post dose
Plasma 3TC Vz/F | 48 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States